CLINICAL TRIAL: NCT02006732
Title: A Randomised, Double-blind, Placebo- and Active-controlled Parallel Group Study to Assess the Efficacy of 12 Weeks of Once Daily Treatment of Two Doses of Orally Inhaled Tiotropium+ Olodaterol Fixed Dose Combination (Delivered by the Respimat Inhaler) in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Tiotropium+Olodaterol Fixed Dose Combination (FDC) in Chronic Obstructive Pulmonary Disease (OTEMTO 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.26; 2013-002264-24 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-10-14; First posted 2013-12-10 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Tiotropium Bromide

ARMS (4):
- tiotropium + olodaterol low dose (Experimental): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: olodaterol; Drug: tiotropium
- tiotropium + olodaterol high dose (Experimental): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: olodaterol; Drug: tiotropium
- tiotropium (Active Comparator): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: tiotropium
- placebo (Placebo Comparator): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: olodaterol — fixed dose combination
  Arms: tiotropium + olodaterol high dose; tiotropium + olodaterol low dose
Drug: tiotropium — fixed dose combination
  Arms: tiotropium; tiotropium + olodaterol high dose; tiotropium + olodaterol low dose
Drug: placebo
  Arms: placebo

SUMMARY:
The objective of this study is to assess the efficacy and safety of 12 weeks once daily treatment with orally inhaled tiotropium + olodaterol FDC (delivered by the Respimat inhaler) compared with tiotropium and placebo in patients with COPD.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis chronic obstructive pulmonary disease
* Relatively stable airway obstruction with post FEV1 >=30 and < 80% predicted normal and post FEV1/ FVC < 70%
* Male or female patients, 40 years of age or more
* Smoking history more than 10 pack years

Exclusion criteria:

* Significant diseases other than COPD
* History of asthma
* COPD exacerbation in previous 3 months
* Completion of pulmonary rehabilitation program within previous 6 weeks or current participation in pulmonary rehabilitation program.
* Pregnant or nursing women
* Patients unable to comply with pulmonary medication restrictions

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 809 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (78):
- United States (20):
  - 1237.26.10620 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1237.26.10618 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1237.26.10619 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1237.26.10614 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1237.26.10616 Boehringer Ingelheim Investigational Site, Duluth, Georgia
  - 1237.26.10613 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1237.26.10615 Boehringer Ingelheim Investigational Site, Greensboro, North Carolina
  - 1237.26.10603 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1237.26.10621 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1237.26.10612 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1237.26.10605 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1237.26.10606 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1237.26.10610 Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - 1237.26.10607 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 1237.26.10617 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1237.26.10608 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1237.26.10604 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1237.26.10609 Boehringer Ingelheim Investigational Site, Boerne, Texas
  - 1237.26.10602 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1237.26.10601 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia
- Australia (6):
  - 1237.26.61004 Boehringer Ingelheim Investigational Site, Concord, New South Wales
  - 1237.26.61002 Boehringer Ingelheim Investigational Site, Daw Park, South Australia
  - 1237.26.61003 Boehringer Ingelheim Investigational Site, Toorak Gardens, South Australia
  - 1237.26.61007 Boehringer Ingelheim Investigational Site, Woodville, South Australia
  - 1237.26.61005 Boehringer Ingelheim Investigational Site, Murdoch, Western Australia
  - 1237.26.61001 Boehringer Ingelheim Investigational Site, Nedlands, Western Australia
- Austria (5):
  - 1237.26.43004 Boehringer Ingelheim Investigational Site, Feldbach
  - 1237.26.43002 Boehringer Ingelheim Investigational Site, Grieskirchen
  - 1237.26.43003 Boehringer Ingelheim Investigational Site, Linz
  - 1237.26.43006 Boehringer Ingelheim Investigational Site, Linz
  - 1237.26.43001 Boehringer Ingelheim Investigational Site, Thalheim bei Wels
- Canada (9):
  - 1237.26.11605 Boehringer Ingelheim Investigational Site, Moncton, New Brunswick
  - 1237.26.11609 Boehringer Ingelheim Investigational Site, Courtice, Ontario
  - 1237.26.11608 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1237.26.11606 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.26.11607 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.26.11601 Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - 1237.26.11611 Boehringer Ingelheim Investigational Site, Mirabel, Quebec
  - 1237.26.11602 Boehringer Ingelheim Investigational Site, Point Claire, Quebec
  - 1237.26.11603 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
- Germany (16):
  - 1237.26.49610 Boehringer Ingelheim Investigational Site, Bamberg
  - 1237.26.49611 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.26.49616 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.26.49609 Boehringer Ingelheim Investigational Site, Bochum
  - 1237.26.49607 Boehringer Ingelheim Investigational Site, Dresden
  - 1237.26.49612 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1237.26.49615 Boehringer Ingelheim Investigational Site, Halberstadt
  - 1237.26.49606 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.26.49608 Boehringer Ingelheim Investigational Site, Hanover
  - 1237.26.49603 Boehringer Ingelheim Investigational Site, Hettstedt
  - 1237.26.49604 Boehringer Ingelheim Investigational Site, Leipzig
  - 1237.26.49605 Boehringer Ingelheim Investigational Site, Leipzig
  - 1237.26.49601 Boehringer Ingelheim Investigational Site, Lübeck
  - 1237.26.49602 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1237.26.49614 Boehringer Ingelheim Investigational Site, Schwerin
  - 1237.26.49613 Boehringer Ingelheim Investigational Site, Wiesloch
- Greece (5):
  - 1237.26.30005 Boehringer Ingelheim Investigational Site, Athens
  - 1237.26.30002 Boehringer Ingelheim Investigational Site, Heraklion
  - 1237.26.30001 Boehringer Ingelheim Investigational Site, Nafplion
  - 1237.26.30004 Boehringer Ingelheim Investigational Site, Serres
  - 1237.26.30003 Boehringer Ingelheim Investigational Site, Thessaloniki
- 1237.26.64001 Boehringer Ingelheim Investigational Site, Greenlane East Auckland NZ, New Zealand
- Norway (4):
  - 1237.26.47003 Boehringer Ingelheim Investigational Site, Hamar
  - 1237.26.47001 Boehringer Ingelheim Investigational Site, Hønefoss
  - 1237.26.47002 Boehringer Ingelheim Investigational Site, Kløfta
  - 1237.26.47004 Boehringer Ingelheim Investigational Site, Lierskogen
- Slovakia (4):
  - 1237.26.42103 Boehringer Ingelheim Investigational Site, Bardejov
  - 1237.26.42104 Boehringer Ingelheim Investigational Site, Humenné
  - 1237.26.42102 Boehringer Ingelheim Investigational Site, Spišská Nová Ves
  - 1237.26.42101 Boehringer Ingelheim Investigational Site, Vyšné Hágy
- South Africa (4):
  - 1237.26.27601 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.26.27602 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.26.27604 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.26.27605 Boehringer Ingelheim Investigational Site, Durban
- Sweden (4):
  - 1237.26.46004 Boehringer Ingelheim Investigational Site, Höllviken
  - 1237.26.46001 Boehringer Ingelheim Investigational Site, Lund
  - 1237.26.46002 Boehringer Ingelheim Investigational Site, Stockholm
  - 1237.26.46003 Boehringer Ingelheim Investigational Site, Uddevalla

REFERENCES:
- [Derived] Buhl R, de la Hoz A, Xue W, Singh D, Ferguson GT. Efficacy of Tiotropium/Olodaterol Compared with Tiotropium as a First-Line Maintenance Treatment in Patients with COPD Who Are Naive to LAMA, LABA and ICS: Pooled Analysis of Four Clinical Trials. Adv Ther. 2020 Oct;37(10):4175-4189. doi: 10.1007/s12325-020-01411-0. Epub 2020 Jul 15. PMID 32671684
- [Derived] Buhl R, Singh D, de la Hoz A, Xue W, Ferguson GT. Benefits of Tiotropium/Olodaterol Compared with Tiotropium in Patients with COPD Receiving only LAMA at Baseline: Pooled Analysis of the TONADO(R) and OTEMTO(R) Studies. Adv Ther. 2020 Aug;37(8):3485-3499. doi: 10.1007/s12325-020-01373-3. Epub 2020 May 27. PMID 32462607
- [Derived] Singh D, Gaga M, Schmidt O, Bjermer L, Gronke L, Voss F, Ferguson GT. Effects of tiotropium + olodaterol versus tiotropium or placebo by COPD disease severity and previous treatment history in the OTEMTO(R) studies. Respir Res. 2016 Jun 18;17(1):73. doi: 10.1186/s12931-016-0387-7. PMID 27316465
- [Derived] Singh D, Ferguson GT, Bolitschek J, Gronke L, Hallmann C, Bennett N, Abrahams R, Schmidt O, Bjermer L. Tiotropium + olodaterol shows clinically meaningful improvements in quality of life. Respir Med. 2015 Oct;109(10):1312-9. doi: 10.1016/j.rmed.2015.08.002. Epub 2015 Aug 12. PMID 26320402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 809 patients were randomised and treated.
Groups:
- Placebo: Once daily 2 puffs solution of placebo for inhalation with Respimat
- Tiotropium 5 μg: Once daily 2 puffs solution of 2.5 μg tiotropium for inhalation with Respimat
- Tiotropium 2.5 μg+ Olodaterol 5 μg: Once daily 2 puffs solution of 1.25 μg tiotropium / 2.5 μg olodaterol for inhalation with Respimat.
- Tiotropium 5 μg + Olodaterol 5 μg: Once daily 2 puffs solution of 2.5 μg tiotropium / 2.5 μg olodaterol for inhalation with Respimat.
Period: Overall Study
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg+ Olodaterol 5 μg | Tiotropium 5 μg + Olodaterol 5 μg
Started | 202 | 203 | 202 | 202
Completed | 182 | 191 | 193 | 198
Not Completed | 20 | 12 | 9 | 4
Not completed — Adverse Event | 10 | 7 | 4 | 2
Not completed — Lack of Efficacy | 6 | 3 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg+ Olodaterol 5 μg | Tiotropium 5 μg + Olodaterol 5 μg | Total
Number analyzed (Participants) | 202 | 203 | 202 | 202 | 809
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.3) | 64.7 (8.4) | 64.4 (8.6) | 65.2 (8.5) | 64.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 73 | 76 | 69 | 303
  Male | 117 | 130 | 126 | 133 | 506

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-3h Response
Description: Forced expiratory volume in one second (FEV1) Area under the curve (AUC) 0-3h was calculated as the area under the FEV1-time curve from 0 to 3h post-dose using the trapezoidal rule, divided by the duration (3h) to report in litres. FEV1 AUC0-3h response was defined as FEV1 AUC0-3h minus baseline FEV1. The adjusted mean and standard error (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; spatial power covariance structure for within-patient errors and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: baseline and 12 weeks
Population: Patients from the Full Analysis Set (FAS): This patient set included all randomized and treated patients who had a baseline and at least one postbaseline measurement for any of the primary efficacy endpoints.
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg+ Olodaterol 5 μg | Tiotropium 5 μg + Olodaterol 5 μg
Number analyzed (Participants) | 199 | 201 | 200 | 200
L | -0.006 (0.014) | 0.188 (0.013) | 0.279 (0.014) | 0.293 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.299, 95% CI 2-sided [0.261 to 0.336], Standard Error of Mean 0.019
Statistical Analysis 2: Comparison: Tiotropium 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.105, 95% CI 2-sided [0.069 to 0.141], Standard Error of Mean 0.019
Statistical Analysis 3: Comparison: Placebo vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.284, 95% CI 2-sided [0.246 to 0.323], Standard Error of Mean 0.020
Statistical Analysis 4: Comparison: Tiotropium 5 μg vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.091, 95% CI 2-sided [0.053 to 0.128], Standard Error of Mean 0.019
Statistical Analysis 5: Comparison: Placebo vs Tiotropium 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.194, 95% CI 2-sided [0.156 to 0.232], Standard Error of Mean 0.019
Statistical Analysis 6: Comparison: Tiotropium 2.5 μg+ Olodaterol 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.4499, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [-0.023 to 0.051], Standard Error of Mean 0.019

2. Primary Outcome: Trough FEV1 Response (Change From Baseline)
Description: Trough FEV1 was defined as the FEV1 value at the end of the dosing interval (24 hours). It was calculated as the mean of the 2 FEV1 measurements performed 23 h and at 23 h 50 min after inhalation of study medication at day 85. Trough FEV1 response was defines as trough FEV1 minus baseline FEV1. The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; spatial power covariance structure for within-patient errors and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: baseline and 12 weeks
Population: Patients from FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg+ Olodaterol 5 μg | Tiotropium 5 μg + Olodaterol 5 μg
Number analyzed (Participants) | 193 | 197 | 200 | 199
L | -0.003 (0.014) | 0.124 (0.013) | 0.166 (0.013) | 0.163 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.166, 95% CI 2-sided [0.129 to 0.203], Standard Error of Mean 0.019
Statistical Analysis 2: Comparison: Tiotropium 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0395, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [0.002 to 0.076], Standard Error of Mean 0.019
Statistical Analysis 3: Comparison: Placebo vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.169, 95% CI 2-sided [0.132 to 0.207], Standard Error of Mean 0.019
Statistical Analysis 4: Comparison: Tiotropium 5 μg vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0269, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.042, 95% CI 2-sided [0.005 to 0.079], Standard Error of Mean 0.019
Statistical Analysis 5: Comparison: Placebo vs Tiotropium 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.127, 95% CI 2-sided [0.090 to 0.165], Standard Error of Mean 0.019
Statistical Analysis 6: Comparison: Tiotropium 2.5 μg+ Olodaterol 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.8669, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.040 to 0.034], Standard Error of Mean 0.019

3. Primary Outcome: St. George's Respiratory Questionnaire (SGRQ) Total Score Based on Data From This Individual Study
Description: The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; spatial power covariance structure for within-patient errors and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: 12 weeks treatment
Population: Patients from FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg+ Olodaterol 5 μg | Tiotropium 5 μg + Olodaterol 5 μg
Number analyzed (Participants) | 184 | 192 | 195 | 197
units on a scale | 42.575 (0.711) | 39.729 (0.694) | 38.909 (0.691) | 38.011 (0.683)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -4.564, 95% CI 2-sided [-6.499 to -2.629], Standard Error of Mean 0.986
Statistical Analysis 2: Comparison: Tiotropium 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0780, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -1.717, 95% CI 2-sided [-3.628 to 0.193], Standard Error of Mean 0.974
Statistical Analysis 3: Comparison: Placebo vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0002, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -3.666, 95% CI 2-sided [-5.611 to -1.721], Standard Error of Mean 0.991
Statistical Analysis 4: Comparison: Tiotropium 5 μg vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p = 0.4028, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -0.820, 95% CI 2-sided [-2.741 to 1.102], Standard Error of Mean 0.979
Statistical Analysis 5: Comparison: Placebo vs Tiotropium 5 μg; Test type: Superiority or Other; p = 0.0042, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -2.846, 95% CI 2-sided [-4.796 to -0.897], Standard Error of Mean 0.993
Statistical Analysis 6: Comparison: Tiotropium 2.5 μg+ Olodaterol 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.3555, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -0.898, 95% CI 2-sided [-2.804 to 1.008], Standard Error of Mean 0.971

4. Primary Outcome: St. George's Respiratory Questionnaire (SGRQ) Total Score Based on Combined Dataset From This Study and the Replicate Study NCT01964352
Description: This endpoint was evaluated after combining the data from this and the replicate study NCT01964352 as specified in the analysis plan. The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
  The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; spatial power covariance structure for within-patient errors and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: 12 weeks treatment
Population: Patients from FAS after combining the data from this and the replicate study NCT01964352
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg+ Olodaterol 5 μg | Tiotropium 5 μg + Olodaterol 5 μg
Number analyzed (Participants) | 370 | 384 | 394 | 393
units on a scale | 42.265 (0.511) | 39.694 (0.498) | 38.419 (0.494) | 37.597 (0.492)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -4.668, 95% CI 2-sided [-6.060 to -3.276], Standard Error of Mean 0.710
Statistical Analysis 2: Comparison: Tiotropium 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0028, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -2.097, 95% CI 2-sided [-3.471 to -0.723], Standard Error of Mean 0.701
Statistical Analysis 3: Comparison: Placebo vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -3.846, 95% CI 2-sided [-5.240 to -2.451], Standard Error of Mean 0.711
Statistical Analysis 4: Comparison: Tiotropium 5 μg vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0696, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -1.274, 95% CI 2-sided [-2.651 to 0.102], Standard Error of Mean 0.702
Statistical Analysis 5: Comparison: Placebo vs Tiotropium 5 μg; Test type: Superiority or Other; p = 0.0003, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -2.571, 95% CI 2-sided [-3.971 to -1.171], Standard Error of Mean 0.714
Statistical Analysis 6: Comparison: Tiotropium 2.5 μg+ Olodaterol 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.2387, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -0.822, 95% CI 2-sided [-2.191 to 0.546], Standard Error of Mean 0.698

5. Secondary Outcome: Trough Forced Vital Capacity (FVC) Response (Change From Baseline)
Description: Trough FVC was defined as the FVC value at the end of the dosing interval (24 hours). It was calculated as the mean of the 2 FVC measurements performed 23 h and at 23 h 50 min after inhalation of study medication at day 85. Trough FVC response was defined as trough FVC minus baseline FVC. The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; spatial power covariance structure for within-patient errors and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: baseline and 12 weeks
Population: Patients from FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg+ Olodaterol 5 μg | Tiotropium 5 μg + Olodaterol 5 μg
Number analyzed (Participants) | 193 | 197 | 200 | 199
L | -0.021 (0.024) | 0.170 (0.023) | 0.284 (0.023) | 0.231 (0.023)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.252, 95% CI 2-sided [0.187 to 0.317], Standard Error of Mean 0.033
Statistical Analysis 2: Comparison: Tiotropium 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0614, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.061, 95% CI 2-sided [-0.003 to 0.125], Standard Error of Mean 0.033
Statistical Analysis 3: Comparison: Placebo vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.305, 95% CI 2-sided [0.240 to 0.370], Standard Error of Mean 0.033
Statistical Analysis 4: Comparison: Tiotropium 5 μg vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0005, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.114, 95% CI 2-sided [0.049 to 0.178], Standard Error of Mean 0.033
Statistical Analysis 5: Comparison: Placebo vs Tiotropium 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.191, 95% CI 2-sided [0.126 to 0.256], Standard Error of Mean 0.033
Statistical Analysis 6: Comparison: Tiotropium 2.5 μg+ Olodaterol 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.1089, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -0.053, 95% CI 2-sided [-0.117 to 0.012], Standard Error of Mean 0.033

6. Secondary Outcome: TDI Focal Score Based on Data From This Individual Study
Description: Mahler Transitional Dyspnoea Index (TDI) focal score was performed to measure the effect of the treatment on patients' dyspnoea.(Rating scale of 3 components - change in functional impairment, change in magnitude of tasks, change in magnitude of efforts. Worst score = -9, best score = +9).
  The adjusted mean (SE) are obtained from fitting an MMRM model including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; spatial power covariance structure for within-patient errors and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: 12 weeks
Population: Patients from FAS
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg+ Olodaterol 5 μg | Tiotropium 5 μg + Olodaterol 5 μg
Number analyzed (Participants) | 183 | 192 | 195 | 197
Units on a scale | 0.337 (0.195) | 0.950 (0.191) | 1.599 (0.189) | 1.531 (0.187)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 1.195, 95% CI 2-sided [0.665 to 1.725], Standard Error of Mean 0.270
Statistical Analysis 2: Comparison: Tiotropium 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0296, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.582, 95% CI 2-sided [0.058 to 1.106], Standard Error of Mean 0.267
Statistical Analysis 3: Comparison: Placebo vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 1.263, 95% CI 2-sided [0.730 to 1.796], Standard Error of Mean 0.272
Statistical Analysis 4: Comparison: Tiotropium 5 μg vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0159, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.650, 95% CI 2-sided [0.122 to 1.178], Standard Error of Mean 0.269
Statistical Analysis 5: Comparison: Placebo vs Tiotropium 5 μg; Test type: Superiority or Other; p = 0.0248, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.613, 95% CI 2-sided [0.078 to 1.148], Standard Error of Mean 0.273
Statistical Analysis 6: Comparison: Tiotropium 2.5 μg+ Olodaterol 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.7984, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -0.068, 95% CI 2-sided [-0.590 to 0.454], Standard Error of Mean 0.266

7. Secondary Outcome: TDI Focal Score Based on Combined Dataset From This Study and the Replicate Study NCT01964352
Description: This endpoint was evaluated after combining the data from this and the replicate study NCT01964352 as specified in the analysis plan. Mahler Transitional Dyspnoea Index (TDI) focal score was performed to measure the effect of the treatment on patients' dyspnoea.(Rating scale of 3 components - change in functional impairment, change in magnitude of tasks, change in magnitude of efforts. Worst score = -9, best score = +9).
  The adjusted mean (SE) are obtained from fitting an MMRM model including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; spatial power covariance structure for within-patient errors and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: 12 weeks
Population: Patients from FAS after combining the data from this and the replicate study NCT01964352
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg+ Olodaterol 5 μg | Tiotropium 5 μg + Olodaterol 5 μg
Number analyzed (Participants) | 370 | 385 | 394 | 393
Units on a scale | 0.111 (0.139) | 1.140 (0.136) | 1.722 (0.134) | 1.734 (0.134)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 1.623, 95% CI 2-sided [1.245 to 2.000], Standard Error of Mean 0.193
Statistical Analysis 2: Comparison: Tiotropium 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0019, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.594, 95% CI 2-sided [0.220 to 0.967], Standard Error of Mean 0.190
Statistical Analysis 3: Comparison: Placebo vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 1.611, 95% CI 2-sided [1.232 to 1.989], Standard Error of Mean 0.193
Statistical Analysis 4: Comparison: Tiotropium 5 μg vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p = 0.0023, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.582, 95% CI 2-sided [0.207 to 0.956], Standard Error of Mean 0.191
Statistical Analysis 5: Comparison: Placebo vs Tiotropium 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 1.029, 95% CI 2-sided [0.649 to 1.410], Standard Error of Mean 0.194
Statistical Analysis 6: Comparison: Tiotropium 2.5 μg+ Olodaterol 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.9494, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.012, 95% CI 2-sided [-0.359 to 0.383], Standard Error of Mean 0.189

8. Secondary Outcome: FVC AUC0-3h Response (Change From Baseline)
Description: The adjusted mean (SE) are obtained from fitting a mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; spatial power covariance structure for within-patient errors and Kenward-Roger approximation of denominator degrees of freedom.
Time Frame: baseline and 12 weeks
Population: Patients from FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg+ Olodaterol 5 μg | Tiotropium 5 μg + Olodaterol 5 μg
Number analyzed (Participants) | 199 | 201 | 200 | 200
L | -0.018 (0.025) | 0.266 (0.023) | 0.436 (0.024) | 0.414 (0.023)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.432, 95% CI 2-sided [0.366 to 0.498], Standard Error of Mean 0.033
Statistical Analysis 2: Comparison: Tiotropium 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.148, 95% CI 2-sided [0.084 to 0.212], Standard Error of Mean 0.033
Statistical Analysis 3: Comparison: Placebo vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.455, 95% CI 2-sided [0.387 to 0.522], Standard Error of Mean 0.034
Statistical Analysis 4: Comparison: Tiotropium 5 μg vs Tiotropium 2.5 μg+ Olodaterol 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.171, 95% CI 2-sided [0.105 to 0.236], Standard Error of Mean 0.034
Statistical Analysis 5: Comparison: Placebo vs Tiotropium 5 μg; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = 0.284, 95% CI 2-sided [0.217 to 0.350], Standard Error of Mean 0.034
Statistical Analysis 6: Comparison: Tiotropium 2.5 μg+ Olodaterol 5 μg vs Tiotropium 5 μg + Olodaterol 5 μg; Test type: Superiority or Other; p = 0.4974, Mixed Effects Model for Repeated Measure; Mean Difference (Final Values) = -0.022, 95% CI 2-sided [-0.087 to 0.042], Standard Error of Mean 0.033

ADVERSE EVENTS:
Time Frame: up to 112 days
Groups:
- Tiotropium 2.5 μg +Olodaterol 5 μg: Once daily 2 puffs solution of 1.25 μg tiotropium / 2.5 μg olodaterol for inhalation with Respimat.
- Tiotropium 5 μg +Olodaterol 5 μg: Once daily 2 puffs solution of 2.5 μg tiotropium / 2.5 μg olodaterol for inhalation with Respimat.
Arm/Group | Placebo | Tiotropium 5 μg | Tiotropium 2.5 μg +Olodaterol 5 μg | Tiotropium 5 μg +Olodaterol 5 μg
Serious Adverse Events (participants affected / at risk) | 4/202 | 12/203 | 4/202 | 6/202
Other Adverse Events (participants affected / at risk) | 34/202 | 15/203 | 25/202 | 14/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=202) | Tiotropium 5 μg (N=203) | Tiotropium 2.5 μg +Olodaterol 5 μg (N=202) | Tiotropium 5 μg +Olodaterol 5 μg (N=202)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=202) | Tiotropium 5 μg (N=203) | Tiotropium 2.5 μg +Olodaterol 5 μg (N=202) | Tiotropium 5 μg +Olodaterol 5 μg (N=202)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 | 7 | 17 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 4 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.